CLINICAL TRIAL: NCT05822648
Title: Evaluating a Brief Type 2 Diabetes Prevention Program With Greater Scalability
Brief Title: Evaluating a Type 2 Diabetes Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Eric Stice, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 68320; P30DK116074 (NIH)
Record Dates: First submitted 2023-03-20; First posted 2023-04-21 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes; PreDiabetes
Keywords: prevention; Type 2 Diabetes; prediabetes; group intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and follow-up assessors will be blinded to condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Project Health will be delivered in six 1-hour group sessions that will be held weekly. In addition, participants will be asked to complete 30 mins of response inhibition and attention trainings once per week between the sessions. This program promotes to retain the gradual lifestyle modification designed to bring energy intake into balance with energy output and the food response inhibition and attention training, but will adapt the dissonance-induction activities to focus on the negative effects of developing T2D in addition to the negative effects of obesity, overeating, and a sedentary lifestyle.
  Interventions: Behavioral: Project Health
- Control (Active Comparator): We selected a T2D management psychoeducational comparison condition. To match Project Health, the educational videos will be delivered in 6 1-hour blocks. The educational group will be instructed to watch videos on nutrition, exercise, and how to maintain general health during the lifespan
  Interventions: Other: Educational Video Control

INTERVENTIONS:
Behavioral: Project Health — Project Health will be delivered in six 1-hour group sessions that will be held weekly. In addition, participants will be asked to complete 30 mins of response inhibition and attention trainings once per week between the sessions. This program promotes to retain the gradual lifestyle modification designed to bring energy intake into balance with energy output and the food response inhibition and attention training, but will adapt the dissonance-induction activities to focus on the negative effects of developing T2D in addition to the negative effects of obesity, overeating, and a sedentary lifestyle.
  Arms: Intervention
Other: Educational Video Control — We selected a T2D management psychoeducational comparison condition. To match Project Health, the educational videos will be delivered in 6 1-hour blocks. The educational group will be instructed to watch videos on nutrition, exercise, and how to maintain general health during the lifespan
  Arms: Control

SUMMARY:
This study aims to test the effectiveness of a Type 2 Diabetes (T2D) prevention program for individuals who have been diagnosed with prediabetes compared to a T2D educational control group. Project health is an obesity prevention program and has produced a 42% to 53% reduction in future onset of overweight/obesity and also produced greater reductions in negative affect compared to assessment-only controls that persisted. Project Health has been adapted to prevent onset of T2D among individuals with prediabetes. The study aims to test the effectiveness of Project Health at reducing BMI, HbA1c levels, increase physical activity and improve glucose control.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 65
2. Overweight (BMI between 25 and 40 kg/m2)
3. Diagnosed with prediabetes, defined as having elevated HbA1c (5.7-6.4%).

Exclusion Criteria:

1. Not between the ages of 18 and 65
2. Not overweight (BMI between 25 and 40 kg/m2)
3. Not diagnosed with prediabetes, defined as having elevated HbA1c (5.7-6.4%).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 30 | 32
Completed | 30 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 32 | 62
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 26 | 29 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 19 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 0 | 2
  White | 11 | 8 | 19
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index (BMI) - Post-Test
Description: BMI will be assessed at post-test to see which intervention produced greater reductions in BMI
Time Frame: post-test (immediately after completion of 6 week intervention)
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 31
kg/m2 | 30.3 (6.6) | 28.8 (5.3)

2. Primary Outcome: Body Mass Index (BMI) - 3-Month Follow-Up
Description: BMI will be assessed at 3-month follow-up to see which intervention produced greater reductions in BMI
Time Frame: 3-month follow-up
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 31
kg/m2 | 30.3 (6.5) | 28.7 (5.5)

3. Primary Outcome: HbA1c at 3-month Follow-up
Description: Participants will complete an HbA1c test at 3-month follow-up to determine their pre-diabetes status
Time Frame: 3-month follow-up
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 31
percent | 5.8 (0.4) | 6 (0.4)

4. Primary Outcome: Fasting Plasma Glucose
Description: Participants will complete a fasting glucose test at 3-month follow-up to determine their pre-diabetes status
Time Frame: 3-month follow-up
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 31
mg/dL | 107 (12) | 108 (13)

5. Primary Outcome: Percent Body Fat - Post-Test
Time Frame: post-test (immediately after completion of 6 week intervention)
Measure: Mean (Standard Deviation); unit: percent body fat
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 31
percent body fat | 39.2 (9.5) | 38.4 (7.8)

6. Primary Outcome: Percent Body Fat - 3-Month Follow-Up
Time Frame: 3-month follow-up
Measure: Mean (Standard Deviation); unit: percent body fat
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 31
percent body fat | 38.3 (9.8) | 37.8 (8.0)

7. Primary Outcome: Percent Lean Body Mass - Post-Test
Time Frame: post-test (immediately after completion of 6 week intervention)
Measure: Mean (Standard Deviation); unit: percent lean mass
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 31
percent lean mass | 60.9 (9.6) | 61.6 (7.8)

8. Primary Outcome: Percent Lean Body Mass - 3-Month Follow-Up
Time Frame: 3-month follow-up
Measure: Mean (Standard Deviation); unit: percent lean mass
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 31
percent lean mass | 61.6 (9.7) | 62.2 (7.9)

ADVERSE EVENTS:
Time Frame: 6-week intervention period plus 3-month follow-up
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 0/30 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT05822648/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT05822648/SAP_001.pdf